CLINICAL TRIAL: NCT04954898
Title: Post-market Evaluation of Clinical Outcomes in China for the TECNIS® Multifocal Toric 1-Piece Intraocular Lens Model Series ZMT
Brief Title: Post-market Evaluation of Clinical Outcomes in China for the TECNIS Model ZMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Surgical Vision, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DIOL-301-CZMT
Record Dates: First submitted 2021-06-29; First posted 2021-07-08 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Lens (Experimental): TECNIS Multifocal Toric 1-piece lens, Model ZMT
  Interventions: Device: Study Lens: TECNIS Multifocal Toric 1-piece lens, Model ZMT

INTERVENTIONS:
Device: Study Lens: TECNIS Multifocal Toric 1-piece lens, Model ZMT — Surgeons will perform standardized, small-incision, cataract surgery and implant the study lenses using a JJSV-validated insertion system qualified for use with TECNIS Multifocal Toric 1-Piece IOL.

SUMMARY:
This is a prospective, multicenter, single-arm, open-label clinical study of the commercially available TECNIS Multifocal Toric 1-Piece IOL. The study will enroll up to 120 subjects from up to 8 sites in China. The subjects will be followed for 12-months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female at least 22 years of age
2. Have a cataract in one or both eyes, with planned phacoemulsification with intraocular lens implantation
3. Regular corneal astigmatism that is planned for correction with an intraocular lens in the study eye(s)
4. Availability, willingness and sufficient cognitive awareness to understand the purpose of the examination procedures and comply with postoperative visits that are required by the study protocol
5. Voluntary participation indicated by the study informed consent form (ICF) signed by the patient or legal guardian.

Exclusion Criteria:

1. Concurrent participation or participation in any other clinical study within 30 days prior to the preoperative visit
2. Ocular disease (other than cataract) that may significantly affect postoperative vision, such as visually significant keratopathy, macular lesions, diabetic retinopathy, chronic or severe uveitis, etc.
3. Planned monovision correction (one eye designated for near correction)
4. Severe or unstable systemic disease that may affect the heart, liver, kidney, lung, endocrine (including thyroid insufficiency), blood, or psychoneurological dysfunction
5. Any other systemic or ocular disease that, in the opinion of the investigator, may affect the patient's eligibility for the study.

   -

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2021-08-11 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
The percentage of eyes that are measured at the 1-day postoperative visit to demonstrate ≤10º change from The intended IOL axis at the end of surgery. | 1 day postoperative
  The axis change is calculated as the absolute difference between intended IOL axis and the axis measured at follow-up visit(s).

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Surgical Vision Clinical Trials, Study Director — Johnson & Johnson Surgical Vision
Locations (7):
- China (7):
  - Xiangya Hospital of Central South University, Kaifu, Changsha
  - Guangzhou Aier Eye Hospital, Guangzhou, Guangdong
  - Daqing Oil Field Central South University, Daqing, Heilongjiang
  - Tianjin Medical University Eye Hospital, Tianjin, Nankai
  - Shanghai Aier Eye Hospital, Xuhui, Shanghai Municipality
  - Shanxi Eye Hospital, Taiyuan, Shanxi
  - Eye Hospital, Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Devices Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA project site at http://yoda.yale.edu
URL: http://yoda.yale.edu